CLINICAL TRIAL: NCT01743664
Title: The Efficacy of Eye Movement Desensitization and Reprocessing (EMDR) in Patients With Post Traumatic Stress Disorder in Multiple Sclerosis. A Randomized Controlled Trial.
Brief Title: The Efficacy of EMDR in Patients With PTSD in Multiple Sclerosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: San Luigi Gonzaga Hospital (Other)
Collaborators: Fondazione Italiana Sclerosi Multipla (Other)
Responsible Party: Principal Investigator, Pier Maria Furlan, Head of the Faculty of Medicine and Surgery San Luigi Gonzaga, San Luigi Gonzaga Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2009/R/11
Record Dates: First submitted 2012-11-21; First posted 2012-12-06 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Posttraumatic Stress Disorders; Multiple Sclerosis
Keywords: Posttraumatic Stress Disorders; Multiple Sclerosis; Eye Movement Desensitization Reprocessing; Psychotherapy; Anxiety; Depression; Quality of Life
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Multiple Sclerosis; Anxiety Disorders; Depression | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eye Movement Desesitization Reprocessing (Experimental): The EMDR protocol follows procedures and phases described by Shapiro (1996). This is a complex treatment that incorporates many different interventions in order to recall trauma-related memories and to subdue them. EMDR processing consists of attending to oscillatory stimulation presented in a visual, auditory or tactile modalities, such as moving the finger from side to side across the patient's visual field or presenting an alternating tapping on the hands alternatively. Eye movements are the most commonly used external stimulus, but if the patient has problems with this kind of stimulation, such as headaches or sensomotor deficits, the therapist chooses tapping as an alternative form of oscillatory stimulation with equivalent therapeutic efficacy.
  Interventions: Behavioral: EMDR
- relaxation (Active Comparator): Relaxation sessions will include diaphragmatic breathing, progressive muscle relaxation, visualisation, and rapid relaxation.
  Interventions: Behavioral: Relaxation

INTERVENTIONS:
Behavioral: EMDR — Patients in the experimental group will undergo 10 weekly sessions of 60 minutes each with EMDR following Shapiro's protocol for traumatic events
  Arms: Eye Movement Desesitization Reprocessing
Behavioral: Relaxation — The patients in the control group will undergo 10 weekly relaxation sessions that include diaphragmatic breathing, progressive muscle relaxation, visualization and rapid relaxation.
  Arms: relaxation

SUMMARY:
Multiple Sclerosis (MS) can be associated to many psychological symptoms. One of the most relevant is the experience of distress related to the disease, that can lead to the development of Post Traumatic Stress Disorder (PTSD). As far as we know there are no studies on the efficacy of psychological treatments in MS in spite of its relevance for patients' quality of life. Primary aim is to evaluate the efficacy of the treatment with Eyes Movement Desensitization and Reprocessing(EMDR) in PTSD secondary to MS. EMDR is the elective treatment (together with Cognitive Behavioural Therapy) for PTSD according to international guidelines. The secondary aims are to evaluate the efficacy of EMDR on the PTSD-associated symptoms of anxiety and depression and Quality of Life. The study design is a randomized clinical trial. Sixty patients with MS and PTSD will be pre-screened by using the IES-R and the Clinician Administered PTSD Scale. The patients will be randomized in two groups (30 in the experimental group and 30 in the control group).The psychological assessment will be performed in both groups with the same timing and tools: at baseline (T0), after treatment (T1) and 6 months later (T2) by two trained clinical psychologists (independent and blind to treatment) with the CAPS and the administration of self reports: Trauma Antecedent Questionnaire, Chicago Multiscale Depression Inventory, Hospital Anxiety and Depression Scale and Functional Assessment of Multiple Sclerosis. The experimental group will undergo 10 weekly sessions of 60 minutes each with EMDR following Shapiro's protocol for traumatic events. The efficacy will be evaluated comparing the results between T0, T1 and T2 and comparing the scores of the experimental and the control groups. Primary outcome measures will be: 1) the proportion of participants at T1 and T2 no longer meeting the Diagnostic and Statistical Manual (DSM IV-TR) diagnostic criteria for PTSD; 2) the reduction of CAPS scores for the four PTSD dimensions from pre-treatment to post-treatment evaluation and follow-up (avoidance, reexperiencing the traumatic event, hyperarousal and numbing). Secondary outcome measures will be: comparison of the scores of CMDI, HADS and FAMS of the two groups at T0, T1 and T2. The statistical procedure applied will be a repeated measures analysis of covariance both on the primary outcome continuous measures and on the secondary ones.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a chronic neurological disease of the Central Nervous System (CNS) that affects both the brain and the spinal cord by destroying the myelin sheath that protects the nerve fibers, leaving plaques or scars on the damaged sites. MS shows a wide range of psychological and psychological-related symptoms, including psychiatric aspects, fatigue and cognitive deficits. In particular, there is a strong evidence of psychiatric disorders associated with MS, the most common being depression, adjustment disorder and anxiety. These occur more frequently at the time of diagnosis communication, during the earlier phases of development of the disease and during relapse episodes. Some studies report a significant association between stressful life-events and relapses, in some cases pointing to frequency and number of stressors as an enhancing factor that can predict a relapsing episode.

The patients may experience distress not only in association with external stressors, but also in relation to the onset or the progression of the disease itself. Diagnosis, relapsing episodes and a worsening of physical functioning may be perceived as traumatic events and may give rise to physiological and emotional posttraumatic symptoms and, in some cases, to Post Traumatic Stress Disorder (PTSD). According to the DSM IV-TR, PTSD is a clinical condition characterised by "the development of characteristic symptoms following exposure to an extreme traumatic stressor involving direct personal experience of an event that involves actual or threatened death or serious injury or other threat to physical integrity. The person's response to the event must involve intense fear, helplessness. The characteristic symptoms resulting from the exposure to the extreme trauma include persistent re-experiencing of the traumatic event, persistent avoidance of stimuli associated with the trauma and numbing of general responsiveness and persistent symptoms of increased arousal. The full symptom picture must be present for more than one month and the disturbance must cause clinically significant distress or impairment in social, occupational or other important areas of functioning" [DSM IV]. Many psychological treatments are available for PTSD, ranging from individual therapy to family therapy and support groups together with interpersonal, relational and psychodynamic psychotherapies; their focus is to desensitise the trauma memory and the meaning of the trauma as well as its power to affect relationships. Among these therapies, the two elective treatments according to international guidelines are the Trauma-focused Cognitive-Behavioural Therapy(CBT-TF) and Eye Movement Desensitisation and Reprocessing (EMDR). CBT-TF focuses on thoughts and beliefs helping people to overcome fear about their painful memories by talking about the trauma repeatedly or by imagining the situation that is realistically safe although still frightening. EMDR is based on the accelerated information processing model integrating elements of different psychotherapies and it is applied through an eight-phase approach. In the EMDR, the patient is induced to focus on his/her negative thoughts, image and body sensation while receiving an "alternate stimulus" (such as eye movements, hand taps or sounds). This procedure leads to desensitisation and emotional reprocessing.

The aims of the study are aim to evaluate whether a treatment based on the EMDR protocol can resolve PTSD or reduce PTS symptoms, also improving the PTS-associated symptoms, such as anxiety and depression. Primary objective : to evaluate the efficacy of the treatment with EMDR on the PTSD in MS. Secondary objectives : To evaluate whether after treatment with EMDR there is an improvement in PTS-associated symptoms of anxiety and depression and an improvement in quality of life.

The recruitment of the patients proceed with a two-step screening: 1) the Impact of Event Scale Revised (IES-R) will be administered to consecutive patients corresponding to the neurological inclusion and exclusion criteria, specifying in the instructions that they consider only the illness as the traumatic event. 2) Patients with scores above the cut off of 33 will be assessed with the SCID in order to confirm diagnosis of PTSD. The research protocol will be proposed to patients with PTSD who meet the inclusion/exclusion criteria, with an explanation of the aims of the study, its relevance for MS patients and the possibility that they may be included, by random assignment, in the treatment or control group for the period of the study, with the same timing and assessment tools. If they agree, they sign the informed consent. Patients will be randomised to the intervention (A) or control (B) group using a block-wise randomisation sequence (block size of 10). Assessment Measures: All patients are evaluated by neurologists with the Expanded Disability Status Scale (EDSS).

The psychological assessment of the patients entering the study will be performed at T0 (baseline evaluation), at T1 (post-treatment evaluation after 12 weeks) and at T2 (follow up evaluation six months later) to determine the reliability of the results.

Measures:

* CLINICIAN ADMINISTERED PTSD SCALE (CAPS): the CAPS is a clinical semi-structured interview based on the DSM IV-TR, which is the gold standard to assess PTSD. It is a 30-item structured interview that meets the DSM IV criteria for PTSD. It assesses 4 dimensions of the PTSD: avoidance, reexperiencing the traumatic event, hyperarousal and numbing. Dissociative symptoms are measured by the three CAPS dissociation items (depersonalization, derealization, and reduction in awareness of one's surroundings). It can be used to make a current (past month) or life-time diagnosis of PTSD or to assess symptoms over the past week.
* TRAUMA ANTECEDENT QUESTIONNAIRE (TAQ): an interview based questionnaire to assess the trauma load due to previous traumas. The TAQ asks for the frequency (never, rarely, commonly) of experiences assigned to 11 domains (ranging from positive experiences like competence and safety, to negative experiences such as neglect, physical, emotional, sexual abuse, and witnessing trauma), separately assess four developmental periods including early childhood (0-6), middle childhood, (7-12), adolescence (13 18), and adults (19+).
* CHICAGO MULTISCALE DEPRESSION INVENTORY (CMDI): the CMDI is a 42-item, self-reporting questionnaire and was developed to assess depression in MS and other chronic diseases. It has three subscales designed to be used either separately or in combination. The mood subscale provides a more conservative indication of depression than total CMDI score and other depression tools.
* HOSPITAL ANXIETY AND DEPRESSION SCALE (HADS): the HADS was developed to identify caseness (possible and probable) of anxiety disorders and depression among patients in non-psychiatric hospital clinics. It is divided into an Anxiety subscale (HADS-A) and a Depression subscale (HADS-D) both containing seven intermingled items . The tool has long been used in studies that involve patients with MS.
* FAMS: Quality of life. The FAMS is a factorially derived self-report scale designed to assess six primary aspects of QOL of patients with MS: Mobility, Symptoms, Emotional Well-Being, General Contentment Thinking and Fatigue, and Family/Social Well- Being.

Treatment: The experimental group will undergo 10 sessions of 60 minutes each of treatment with the EMDR protocol. The EMDR treatment will be conducted by 3 expert psychotherapists with more than 6 years experience in the liaison setting, in possession of II level training degree in EMDR. Relaxation techniques (RT) will be performed by three psychotherapists working in the same facility. Treatments will be independent and blinded from the clinical psychologists conducting the clinical assessments.

The EMDR protocol follows procedures and phases described by Shapiro (1996). This is a complex treatment that incorporates many different interventions in order to recall trauma-related memories and to subdue them. EMDR processing consists of attending to oscillatory stimulation presented in a visual, auditory or tactile modalities, such as moving the finger from side to side across the patient's visual field or presenting an alternating tapping on the hands alternatively. Eye movements are the most commonly used external stimulus, but if the patient has problems with this kind of stimulation, such as headaches or sensomotor deficits, the therapist chooses tapping as an alternative form of oscillatory stimulation with equivalent therapeutic efficacy. Relaxation sessions will follow the same structure as the EMDR sessions, including diaphragmatic breathing, progressive muscle relaxation, visualisation, cue-controlled relaxation, and rapid relaxation.

The efficacy of the EMDR treatment will be evaluated by comparing the results of the tools (CAPS, CMDI, HADS, FAMS) administered to the treated group at T0, T1 and T2 and by comparing the scores of the experimental group with those of the control group. Primary outcome measures will include 1) Proportion of participants at T1 and T2 no longer meeting the DSM IV-TR diagnostic criteria for PTSD (SCID) among patients of the experimental group in comparison with those of the control group; 2) the reduction of CAPS scores for the four PTSD dimensions from pre-treatment to follow-up in both groups (avoidance, re-experiencing the traumatic event, hyperarousal and numbing).

3) Reduction in the IES scores. Scores for anxiety, depression and quality of life will be included as secondary outcome. Dissociative symptoms will be evaluated through the three CAPS dissociation items (Taylor et al., 2003).

Additional expected results: the large number of patients assessed for post traumatic symptoms might improve knowledge both of their prevalence and also of the trauma underlying MS. Even if it is not the primary aim of the study, assessment of the trauma load through the interview-based TAQ will lead to life-trauma evaluation which may be studied for their correlation with the onset of the disease and its emotional correlates. Moreover, in EMDR, associated traumas are defined and treated: given that sessions are video-recorded, their analysis (beyond the three sessions that will be reviewed for treatment fidelity) may add knowledge to the role of the trauma load in MS.

ELIGIBILITY:
Inclusion Criteria:

* definite diagnosis of MS (Mc Donald Criteria) evaluated by a neurologist at least six months previously;
* a relapsing-remitting, primary or secondary progressive disease;
* clinically inactive phase of the disease;
* fluent Italian speaker;
* legal capacity to consent to the treatment;
* diagnosis of PTSD assessed with the SCID;
* willingness to suspend all concomitant psychological treatment and suspension of all psychotropic medications at least one month before the treatment or maintenance at baseline level throughout the study.

Exclusion Criteria:

* other serious mental disorders, including bipolar disorders, psychotic symptoms, substance abuse, suicidal tendency or cognitive impairment;
* in corticosteroid treatment during the previous month;
* with other serious medical disorders in addition to MS.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2010-05; Primary Completion 2013-03 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants no longer meeting the DSM IV-TR diagnostic criteria for PTSD among patients of the experimental group in comparison with those of the control group after the treatment. | Change from Baseline of number of patients meeting the PTSD DSM IV-TR criteria at 3 months

SECONDARY OUTCOMES:
Reduction in the IES scores after the treatment. | Reduction from Baseline of IES-R score at 3 months
Proportion of participants no longer meeting the DSM IV-TR diagnostic criteria for PTSD among patients of the experimental group in comparison with those of the control group at the follow up. | Change from Baseline of number of patients meeting the PTSD DSM IV-TR criteria at 9 months
Reduction in the IES scores at the follow-up. | Reduction from Baseline of IES-R score at 9 months

OTHER OUTCOMES:
Reduction of PTS-associated symptoms of anxiety and depression and an improvement in quality of life after the treatment. | Reduction from baseline of PTS-associated symptoms of anxiety and depression and an improvement in quality of life at 3 months.
Reduction of PTS-associated symptoms of anxiety and depression and an improvement in quality of life at the follow-up. | Reduction from baseline of PTS-associated symptoms of anxiety and depression and an improvement in quality of life at 9 months.

CONTACTS AND LOCATIONS:
Overall Officials: Pier M Furlan, M.D., Principal Investigator — San Luigi Gonzaga University Hospital
Locations (1):
- San Luigi Gonzaga University Hospital, Orbassano, Torino, Italy

REFERENCES:
- [Background] Chalfant AM, Bryant RA, Fulcher G. Posttraumatic stress disorder following diagnosis of multiple sclerosis. J Trauma Stress. 2004 Oct;17(5):423-8. doi: 10.1023/B:JOTS.0000048955.65891.4c. PMID 15633921
- [Background] Bisson JI, Ehlers A, Matthews R, Pilling S, Richards D, Turner S. Psychological treatments for chronic post-traumatic stress disorder. Systematic review and meta-analysis. Br J Psychiatry. 2007 Feb;190:97-104. doi: 10.1192/bjp.bp.106.021402. PMID 17267924
- [Background] Kangas M, Henry JL, Bryant RA. Posttraumatic stress disorder following cancer. A conceptual and empirical review. Clin Psychol Rev. 2002 May;22(4):499-524. doi: 10.1016/s0272-7358(01)00118-0. PMID 12094509
- [Background] Tedstone JE, Tarrier N. Posttraumatic stress disorder following medical illness and treatment. Clin Psychol Rev. 2003 May;23(3):409-48. doi: 10.1016/s0272-7358(03)00031-x. PMID 12729679
- [Result] Ostacoli L, Carletto S, Borghi M, Cavallo M, Rocci E, Zuffranieri M, Malucchi S, Bertolotto A, Zennaro A, Furlan PM, Picci RL. Prevalence and significant determinants of post-traumatic stress disorder in a large sample of patients with multiple sclerosis. J Clin Psychol Med Settings. 2013 Jun;20(2):240-6. doi: 10.1007/s10880-012-9323-2. PMID 23053829
- [Derived] Carletto S, Borghi M, Bertino G, Oliva F, Cavallo M, Hofmann A, Zennaro A, Malucchi S, Ostacoli L. Treating Post-traumatic Stress Disorder in Patients with Multiple Sclerosis: A Randomized Controlled Trial Comparing the Efficacy of Eye Movement Desensitization and Reprocessing and Relaxation Therapy. Front Psychol. 2016 Apr 21;7:526. doi: 10.3389/fpsyg.2016.00526. eCollection 2016. PMID 27148134
- See also: link to the Italian Association of Multiple Sclerosis and to its Research Foundation — http://www.aism.it/index.aspx?codpage=ricerca_finanziata